CLINICAL TRIAL: NCT03426059
Title: Mapping the Phenotype in Adults With Phelan-McDermid Syndrome
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Phelan-McDermid Syndrome Foundation (Other)
Responsible Party: Principal Investigator, Mustafa Sahin, Assistant in Neurology, Associate Professor of Neurology, Harvard Medical School, Boston Children's Hospital
Other Study IDs: IRB-P00025776
Record Dates: First submitted 2018-01-31; First posted 2018-02-08 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Phelan-McDermid Syndrome; Autism Spectrum Disorder; Intellectual Disability
Keywords: Phelan-McDermid Syndrome; PMS; Genotype; Phenotype; Mapping; 22q13 Deletion Syndrome; SHANK3; Autism Spectrum Disorder; ASD; Intellectual Disability; ID
MeSH Terms: conditions — Telomeric 22q13 Monosomy Syndrome; Autism Spectrum Disorder; Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draw or saliva sample for future correlative studies in the PMS Biorepository of the Developmental Synaptopathies Consortium
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Phelan-McDermid Syndrome: Phelan-McDermid Syndrome
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention. This is an observational study.

SUMMARY:
The protocol aims to comprehensively define the phenotype of Phelan-McDermid Syndrome and to identify potential genetic factors, which may play a role in the variability of the disease's outcomes. The first aim involves a physical exam, a neurological exam, collection of medical history information, a clinical genetic evaluation, blood work and neuropsychological assessments. If clinically indicated, the protocol collects information from medical tests. These medical tests may include electrocardiography, echocardiography, renal ultrasonography, and renal ultrasound.

DETAILED DESCRIPTION:
Phelan-McDermid syndrome (PMS) or 22q13 Deletion syndrome, caused by a loss of one copy of the SHANK3 gene, is characterized by global developmental delay/intellectual disability, motor skills deficits, delayed or absent speech, and autism spectrum disorder. The goal of this study is to understand more about the PMS phenotypic outcomes and the biological pathways associated in the disorder, and to establish the foundation for future clinical trials in PMS and in other ID/ASD-associated disorders that share signaling pathways with PMS.

Individuals with PMS will be asked to participate in this study if they are 22 years of age or older with pathogenic deletions or mutations of the SHANK3 gene at time of enrollment. Both males and females will be asked to participate. Additionally, to be eligible for study participation, individuals' primary communicative language must be English. Parents and unaffected siblings may also be asked to consent to have blood drawn for analysis.

For this study, there is only one study visit. Study visit involves a physical exam, medical history questions, blood work and neuropsychological assessments. Individuals who have certain clinically indicated procedures (i.e. MRI, EEG, etc.) due will have them done as part of the research study

ELIGIBILITY:
Inclusion Criteria:

* Participant is 22 years of age and older at the time of enrollment
* Participant has been diagnosed with pathogenic deletions or mutations of the SHANK3 gene
* Participant is proficient in English
* Participant provided consent

Exclusion Criteria:

* None

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 adult subjects with PMS will be enrolled across the 6 sites for this study
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Global cognitive ability | Baseline
  Using standardized T-scores from the Mullen Scales for Early Learning (49 to 155, where higher values represent a better outcome) or full scale IQ scores from the Stanford Binet-5 (40 to 160, where higher values represent a better outcome) to measure global cognitive ability
Measure of Adaptive Behavior | Baseline
  Using the standardized composite score from the Vineland Adaptive Behavior Scales (20-160, where higher values represent a better outcome) to measure adaptive behavior
Measure of Overall Language Abilities | Baseline
  Using standardized T-scores from the Mullen Receptive Language and Expressive Language subscales (20 to 80, where higher values represent a better outcome), the standardized composite score Vineland Communication subscale (20-160, where higher values represent a better outcome) and the total raw scores from the Macarthur Bates Communication Developmental Inventory to measure overall language
Measure of Overall Motor Functioning | Baseline
  Using standardized T-scores from the Mullen Gross and Fine Motor subscales (20-80, where higher values represent a better outcome) and the Vineland's Motor Skills Domain Standard Score (20-160, where higher values represent a better outcome) to assess motor ability
Measure of autism symptoms | Baseline
  Using the standardized comparison score from the Autism Diagnostic Observation Scale (1-10, where higher values represent a worse outcome) to measure autism

SECONDARY OUTCOMES:
Measure of Receptive Language Abilities | Baseline
  Using standardized scores from the Peabody Picture Vocabulary Test (20-160, where higher values represent a better outcome) to measure receptive language abilities
Measure of Expressive Language Abilities | Baseline
  Using standardized scores from the Expressive Vocabulary Test (20-160, where higher values represent a better outcome) to measure expressive language abilities

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kolevzon, MD, Study Chair — Seaver Autism Center, Mount Sinai School of Medicine
Locations (6):
- United States (6):
  - Stanford University, Stanford, California
  - Rush University Medical Center, Chicago, Illinois
  - National Institutes of Health, Bethesda, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Texas Southwestern, Dallas, Texas